CLINICAL TRIAL: NCT04871360
Title: Effect of Oral L-Citrulline Supplementation on Liver Function and Non-Alcoholic Fatty Liver Disease in Adolescents With Obesity
Brief Title: Effect of L-Citrulline Supplementation on NAFLD in Adolescents With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Ma Eugenia Garay Sevilla, Titular Research Professor, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAFLD-CITRULLINE
Record Dates: First submitted 2021-04-25; First posted 2021-05-04 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity
Keywords: NAFLD; Obesity; Adolescents; L-citrulline supplementation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Intervention Model Description: The intervention consists of the oral administration of placebo or l-citrulline as follows:
  Group Placebo: Carboxymethyl cellulose will be used for the placebo group. Four capsules will be taken in the morning before the first meal and four capsules at night before going to sleep for eight weeks.
  Group Citrulline: a dose of 6 g of citrulline will be used per day, distributed as 3 g (4 capsules) in the morning before the first meal and 3 g (4 capsules) in the evening before sleep, for eight weeks. Each capsule contains 750 mg of pure citrulline.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The selection of which group each adolescent will belong to will be made by randomization by simple lottery by a researcher from the Department of Medical Sciences of the University of Guanajuato who is not involved in the treatment and follow-up of the participants and will be designated to a Placebo group and to the Citrulline group. The participants and the researcher will not know which group each adolescent belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citrulline group (Experimental): Group of adolescents supplemented orally with 6 g / day of pure L-citrulline in capsules. The dose will be met by taking four (3 g) capsules in the morning before the first meal and four capsules (3 g) in the evening after the last meal.
  Interventions: Dietary Supplement: L-Citrulline supplement
- Placebo group (Placebo Comparator): Group of adolescents supplemented with placebo (carboxymethyl cellulose). The indication for taking will be the same as in the experimental group, four capsules in the morning before the first meal and four capsules at night, after the last meal.
  Interventions: Dietary Supplement: Carboxymethyl cellulose supplement

INTERVENTIONS:
Dietary Supplement: L-Citrulline supplement — The intervention will consist of oral supplementation of six grams of pure l-citrulline for eight weeks.
  Arms: Citrulline group
Dietary Supplement: Carboxymethyl cellulose supplement — The intervention will consist of oral carboxymethyl cellulose supplementation as a placebo.
  Arms: Placebo group

SUMMARY:
One of the comorbidities of obesity is nonalcoholic fatty liver disease (NAFLD). L-citrulline is a non-protein amino acid that has shown positive effects on the degree of fat retention and metabolic profile in NAFLD. The objective is to assess the effect of oral L-citrulline supplementation on liver function and nonalcoholic fatty liver in adolescents with obesity. A clinical study will be carried out in 40 adolescents (15-19 years) with obesity, they will be divided into a control group that will receive a placebo and an experimental group that will receive 6 g of l-citrulline per day for eight weeks.

DETAILED DESCRIPTION:
It is hypothesized that l-citrulline supplementation decreases liver enzymes and the degree of hepatic steatosis in adolescents with obesity. The aim of the study is to assess the effect of oral L-citrulline supplementation on liver function and nonalcoholic fatty liver in adolescents with obesity. A prospective randomized, double-blind clinical study will be carried out in 40 adolescents (15-19 years) with obesity, they will be divided into a control group that will receive a placebo (carboxymethyl cellulose) and an experimental group that will receive 6 g of pure l-citrulline per day per eight weeks. At the beginning and end of the intervention, anthropometric, biochemical and metabolic data will be evaluated, as well as tests of function and degree of hepatic steatosis.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 15 and 19 years old, residents of the city of León, Guanajuato, with obesity due to BMI ≥30 kg / m2 equivalent to the categorization of adults. That they are in stage 5 of Tanner scale with diagnosis of mild, moderate or severe NAFLD and / or alterations in liver enzyme levels. Not be under nutritional treatment, not be smokers, not taking multivitamins, if so, a wash time of 30 days will be given. Not be allergic to l-citrulline or watermelon. Alcohol consumption less than 21 standard drink units for men and 14 standard drink units for women per week (Standard drink: any drink with more than 14 g of pure alcohol).

Exclusion Criteria:

* Present intolerance to l-citrulline or allergy to watermelon.
* Have an adherence of less than 80 percent of the treatments.
* Present other causes of liver disease.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Degree of hepatic steatosis | Baseline to 8 weeks
  The degree of hepatic steatosis will be evaluated by abdominal ultrasound. It will be diagnosed as:
  1. Mild, when an increase in echogenicity and hepatomegaly are observed.
  2. Moderate, when sound attenuation is added.
  3. Severe, when the wall of the portal vessels and the diaphragm are not visible.

SECONDARY OUTCOMES:
Glucose | Baseline to 8 weeks
  Glucose will be evaluated by the GOD-PAD Lakeside glucose oxidase method.
Insulin | Baseline to 8 weeks
  The insulin level will be measured by ELISA (ALPCO) method. The HOMA-IR index will be calculated to determine insulin resistance.
Insulin resistance | Baseline to 8 weeks
  The HOMA-IR index to determine insulin resistance will be calculated from serum glucose and insulin levels.
Lipid profile | Baseline to 8 weeks
  The lipid profile will be measured by the modified Huang method of the Spinreact brand.
LDL-cholesterol | Baseline to 8 weeks
  LDL-cholesterol will be determined using the Friedwald formula.
Urea levels | Baseline to 8 weeks
  Urea levels will be obtained by the Urease GLDH kinetic method.
Uric acid levels | Baseline to 8 weeks
  Uric acid will be evaluated by peroxidase enzymes and colorimetry.
Liver function | Baseline to 8 weeks
  Liver function will be evaluated using the liver enzymes alanine aminotransferase and aspartate aminotransferase by the UV enzymatic kinetic method, as well as with alkaline phosphatase by the optimized kinetic method and direct bilirubin by the DMSO method (dimethyl sulfoxide-Malloy-Evelyn reaction).

CONTACTS AND LOCATIONS:
Overall Officials: Ma. E Garay-Sevilla, PhD, Principal Investigator — Universidad de Guanajuato; Verónica I Tovar-Villegass, Bachelor, Study Chair — Universidad de Guanajuato
Locations (1):
- University of Guanajuato, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No
At the request of the researcher.